CLINICAL TRIAL: NCT02645435
Title: Consequence of the Learning Curve in Direct Anterior Approach for Total Hip Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera Bolognini di Seriate Bergamo (Other)
Responsible Party: Principal Investigator, Riccardo Compagnoni, Medical Doctor, Azienda Ospedaliera Bolognini di Seriate Bergamo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AObolognini1
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Arthropathy of Hip; Surgery
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hip direct anterior approach (Active Comparator): Patients with hip arthritis
  Interventions: Procedure: hip replacement
- Lateral hip approach (Active Comparator): Patients with hip arthritis
  Interventions: Procedure: hip replacement

INTERVENTIONS:
Procedure: hip replacement — Total hip replacement

SUMMARY:
Background:

Direct anterior approach to the hip (DAA) is being considered as one of the most promising minimally-invasive approaches in total hip arthroplasty (THA). Purpose of this study is to analyse influence of learning curve on clinical and radiographic outcome in direct anterior approach (DAA) for total hip replacement.

Methods:

The first 30 patients operated with DAA (group B) were compared to 39 patients operated by Hardinge approach (group A). Peri-and postoperative complications, Harris Hip Score (HHS), implant positioning, experienced pain and patient satisfaction were evaluated at a mean follow-up of 32 months.

DETAILED DESCRIPTION:
Direct anterior approach to the hip (DAA) is being considered as one of the most promising minimally-invasive approaches in total hip arthroplasty (THA). Purpose of this study is to analyse influence of learning curve on clinical and radiographic outcome in direct anterior approach (DAA) for total hip replacement.

Methods:

The first 30 patients operated with DAA (group B) were compared to 39 patients operated by Hardinge approach (group A). Peri-and postoperative complications, Harris Hip Score (HHS), implant positioning, experienced pain and patient satisfaction were evaluated at a mean follow-up of 32 months.

ELIGIBILITY:
Inclusion Criteria:

* Hip arthritis

Exclusion Criteria:

* BMI>35

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical outcome of direct hip approach | 32 months
  Harry's hip score, a clinical score used in orthopedic surgery to describe outcome of hip function

SECONDARY OUTCOMES:
radiological positioning of cup in the replaced hip | 32 months
  using standard x-ray of the hip placement of implants is measured in angles between the iliac line and component line for the cup
radiological positioning of the stem in replaced hip | 32 months
  using standard x-ray of the hip placement of implants is measured in angles between the axis of implant and femoral axis